CLINICAL TRIAL: NCT05052840
Title: Effects of Back Muscles Endurance Training on Pain, Disability, Endurance and Lumbar Flexibility in Patients With Chronic Mechanical Low Back Pain
Brief Title: Effects of Back Muscles Endurance Training in Patients With Chronic Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/0125 Faraz
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Mechanical Low Back Pain; Paraspinal Muscles; Muscle Stretching Exercises
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle endurance training (MET) (Experimental)
  Interventions: Other: Muscle endurance training (MET); Other: Conventional Treatment
- Conventional Treatment (Active Comparator)
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Muscle endurance training (MET) — Experimental group will be given MET Program, stretching & strengthening exercises and Hot packs (for 15 minutes). MET program will include warm up, endurance and cool down exercises. The warm up and cool down period will be consisted of 5-minute walking, and 10 repetitions of stretching exercises. Endurance exercises will consist of 4 levels.
  Arms: Muscle endurance training (MET)
Other: Conventional Treatment — Conventional treatment group will be given hot packs (for 15 minutes) and Strengthening & stretching exercise program including:
  STRETCHING EXERCISES (lumbar extensor muscles, iliopsoas muscles, hamstring muscles, gastrocnemius muscles and pectoral muscles).
  STRENGTHENING EXERCISES (rectus abdominus crunch, oblique crunch, pelvic elevation, single leg pelvic elevation, lumbal spine extension, on hands and knees position with the raise of one leg, on hands and knees position with the raise of opposite arm and leg). Each exercise will be repeated 10 times.

SUMMARY:
Low back pain is one the leading cause of disability and affecting many individuals. Chronic low back pain is associated with restriction in daily physical activities that ultimately leads to disuse atrophy of muscles. The objective of the study is to find out the effects of Back Muscles Endurance Training on pain, disability, endurance and Lumbar flexibility in patients with chronic mechanical low back pain.

DETAILED DESCRIPTION:
Low back pain is the leading worldwide cause of years lost to disability and its burden is growing alongside the increasing and ageing population. Mechanical low back pain refers to back pain that arises intrinsically from the spine, intervertebral disks, or surrounding soft tissues. Repetitive trauma and overuse are common causes of chronic mechanical low back pain, which is often secondary to workplace injury. Most patients who experience activity-limiting low back pain go on to have recurrent episodes. Low back pain is a common condition affecting many individuals at some point in their lives. Chronic low back pain prevalence increases linearly from the third decade of life on, until the 60 years of age, being more prevalent in women.

ELIGIBILITY:
Inclusion Criteria:

* The ages between 20-45 years
* Both Males and Females
* The presence of low back pain as a primary complaint
* The onset of pain at least three months back

Exclusion Criteria:

* Tumors, infection or inflammatory diseases affecting the spine
* Spinal or lower limb surgery
* Spinal fractures or structural deformities such as spinal stenosis, spondylolisthesis and spondylolysis
* Signs of nerve root compression
* Any contraindications for exercise therapy
* Patient with any spinal surgery, have respiratory or systemic diseases.
* Pregnant women.
* Sacroiliac joint dysfunction (determined by any three positives among distraction test, Gaenslen's test, Thigh thrust test, Sacral thrust test, and compression test)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE | 6 weeks
  NPRS is anchored by terms describing pain severity extremes. The 11-point numeric with 0 representing No pain, 1-3 representing Mild Pain (nagging, annoying, interfering little with ADLs), 4-6 representing Moderate Pains (interferes significantly with ADLs), 7-10 representing Sever Pain (disabling, unable to perform ADLs)
REVISED OSWESTERY DISABILITY INDEX (RODQ) | 6 weeks
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. This scale contain question related to functional activities of pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. For patients understanding, URDU version is used.
PRONE DOUBLE STRAIGHT-LEG RAISE TEST | 6 weeks
  The prone double straight-leg raise test will be used to assess participants' back muscle endurance. The participant lay on the plinth in prone-lying position, hips extended, with the hands underneath the forehead and the arms perpendicular to the body. Instruct the participant to raise both legs until knee clearance is achieved. The researcher will monitoring knee clearance by sliding one hand under the thighs. The time taken by participant to maintain knee clearance monitored with a stopwatch will be recorded in seconds as back muscle endurance
MODIFIED SCHOBER'S TEST | 6 weeks
  The patient is standing with his back towards the examiner. The examiner determines the location of the lumbosacral junction at the level of the posterior superior iliac spine by pressing the location of the dimples of Venus. The intersection of the top of the dimples of Venus is marked by drawing a horizontal line. This line acts as the landmark. Two other marks will be drawn 10 cm above and 5 cm below the first landmark. The patient will then be asked to bend over and touch his or her toes as long as possible without increasing pain. The examiner will measure the increase in distance between the superior and inferior marks. The length increment, which is the difference between the 15-cm distance (neutral position) and the increased distance (anterior flexion posture), will be calculated to determine the range of motion of the lumbar spine

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Zohra Shafi Free Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchbinder R, van Tulder M, Oberg B, Costa LM, Woolf A, Schoene M, Croft P; Lancet Low Back Pain Series Working Group. Low back pain: a call for action. Lancet. 2018 Jun 9;391(10137):2384-2388. doi: 10.1016/S0140-6736(18)30488-4. Epub 2018 Mar 21. PMID 29573871
- [Background] Will JS, Bury DC, Miller JA. Mechanical Low Back Pain. Am Fam Physician. 2018 Oct 1;98(7):421-428. PMID 30252425
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Akhtar MW, Karimi H, Gilani SA. Effectiveness of core stabilization exercises and routine exercise therapy in management of pain in chronic non-specific low back pain: A randomized controlled clinical trial. Pak J Med Sci. 2017 Jul-Aug;33(4):1002-1006. doi: 10.12669/pjms.334.12664. PMID 29067082
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Rigoard P, Blond S, David R, Mertens P. Pathophysiological characterisation of back pain generators in failed back surgery syndrome (part B). Neurochirurgie. 2015 Mar;61 Suppl 1:S35-44. doi: 10.1016/j.neuchi.2014.10.104. Epub 2014 Nov 20. PMID 25456443
- [Background] Allegri M, Montella S, Salici F, Valente A, Marchesini M, Compagnone C, Baciarello M, Manferdini ME, Fanelli G. Mechanisms of low back pain: a guide for diagnosis and therapy. F1000Res. 2016 Jun 28;5:F1000 Faculty Rev-1530. doi: 10.12688/f1000research.8105.2. eCollection 2016. PMID 27408698
- [Background] Emami F, Yoosefinejad AK, Razeghi M. Correlations between core muscle geometry, pain intensity, functional disability and postural balance in patients with nonspecific mechanical low back pain. Med Eng Phys. 2018 Oct;60:39-46. doi: 10.1016/j.medengphy.2018.07.006. Epub 2018 Aug 1. PMID 30077486
- [Background] Shiri R, Coggon D, Falah-Hassani K. Exercise for the Prevention of Low Back Pain: Systematic Review and Meta-Analysis of Controlled Trials. Am J Epidemiol. 2018 May 1;187(5):1093-1101. doi: 10.1093/aje/kwx337. PMID 29053873